CLINICAL TRIAL: NCT01420328
Title: To Study the Effect of Vytorin on Intracellular Lipid and Inflammation in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Kaleida Health (Other)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MED7120311A
Record Dates: First submitted 2011-05-26; First posted 2011-08-19 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Obese subjects treated with placebo for 6 weeks
  Interventions: Drug: Placebo
- Vytorin Arm (Active Comparator): Obese subjects treated with Vytorin for 6 weeks
  Interventions: Drug: Vytorin

INTERVENTIONS:
Drug: Vytorin — Simvastatin 40 mg and Ezetimibe 10 mg daily combination pill (Vytorin) for 6 weeks
  Other Names: Ezetimibi/Simvastatin 10/40
  Arms: Vytorin Arm
Drug: Placebo — Placebo treatment for 6 weeks
  Other Names: Placebo for Vytorin
  Arms: Placebo Arm

SUMMARY:
This study focuses on the use of Vytorin to study inflammatory markers in subjects with normal cholesterol.

DETAILED DESCRIPTION:
Following the first demonstration by our group that macronutrient (glucose, cream and a high fat high carbohydrate meal) intake results in increased ROS generation and oxidative stress at the cellular and molecular level, the investigators have now shown in our preliminary data that cream intake induces comprehensive inflammation as reflected in increased intranuclear NFkB binding, decreased IkBα expression, increased expression of IL-1β, IL-12, TNFα and other pro-inflammatory mediators. While carrying out these experiments, the investigators asked whether cream intake was associated with an uptake of lipid by peripheral blood mononuclear cells (MNC). Indeed, there was a significant increase in intracellular lipid which was visualized as intracellular lipid droplets. The increase in intracellular lipid droplets was associated with an increase in intracellular superoxide generation; the expression of CD68, a marker for macrophages; and PECAM, the adhesion molecule which mediates trans- endothelial transfer of leucocytes. The investigators also found that the lipid fractions to increase were cholesterol ester, triglyceride and fatty acids. In view of the tantalizing observation that the lipid droplet laden MNC appeared to be monocytes, looked like foam cells and the fact that CD68 expression had increased, there is a possibility that foam cells may be formed in peripheral circulation by monocytes after a lipid rich meal. This simple model of foam cell formation also lends itself for the study of the effect of various lipid lowering drugs. Our investigation will be the first to study this novel paradigm. The investigators plan to study the effect of a cholesterol lowering agent, Vytorin (simvastatin and ezetimibe), on intracellular lipid in MNC, expression of CD68 and PECAM, ROS generation and inflammation in obese subjects. This investigation may provide an additional mechanism of action by which these drugs may reduce atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65years.
2. Obese BMI >30kg/m2
3. LDL cholesterol >100 mg/dl
4. Written and informed consent signed and dated 5. Not on any vitamin/antioxidants

Exclusion Criteria:

1. On any antilipid agents.
2. Triglyceride >500mg/dl
3. Myocardial infarction, angioplasty/stent placement or coronary artery bypass surgery in the past 6 months
4. Patient on chronic use of non-steroidal anti-inflammatory drugs or steroids
5. Hepatic disease
6. Renal impairment
7. History of drug or alcohol abuse
8. Participation in any other concurrent clinical trial
9. Use of an investigational agent or therapeutic regimen within 30 days of study.
10. Smoker
11. Pregnancy
12. Premenopausal women who are not on birth control pills and have not had a hysterectomy or tubal ligation 13. Anemia with hemoglobin <12 g/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — University at Buffalo, NY
Locations (1):
- Diabetes Endocrinology Center of WNY, Buffalo, New York, United States

REFERENCES:
- [Derived] Ghanim H, Green K, Abuaysheh S, Patel R, Batra M, Chaudhuri A, Makdissi A, Kuhadiya ND, Dandona P. Ezetimibe and simvastatin combination inhibits and reverses the pro-inflammatory and pro-atherogenic effects of cream in obese patients. Atherosclerosis. 2017 Aug;263:278-286. doi: 10.1016/j.atherosclerosis.2017.06.010. Epub 2017 Jun 7. PMID 28711708

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Arm: Placebo tablets given to 10 subjects with obesity but not diabetes and LDL >100 mg/dl on no lipid lowering therapy for a 6 weeks period
- Vytorin Arm: Vytorin: Simvastatin 40 mg and Ezetimibe 10 mg daily combination pill (Vytorin) given to 10 subjects with obesity but not diabetes and LDL >100 mg/dl on no lipid lowering therapy for a 6 weeks period
Period: Overall Study
Arm/Group | Placebo Arm | Vytorin Arm
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Arm/Description: 10 subjects with obesity but not diabetes and LDL >100 mg/dl on placebo treatment for 6 weeks
- Vytorin Arm/Description: 10 subjects with obesity but not diabetes and LDL >100 mg/dl on Vytorin for 6 weeks
  Vytorin: Simvastatin 40 mg and Ezetimibe 10 mg daily combination pill (
- Total: Total of all reporting groups
Arm/Group | Placebo Arm/Description | Vytorin Arm/Description | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at baseline
  years | 49 (4) | 51 (3) | 50 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — United States Of America
  participants
    United States | 10 | 10 | 20
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index
  Kg/m^2 | 38.1 (1.6) | 38.2 (1.7) | 38.2 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in CD68 mRNA Expression in MNC
Description: Percent change from baseline (0 week) in cream challenge induced change in CD68 mRNA expression in MNC after 6 weeks of treatment with Vytorin or placebo.
  Outcome calculated as: (change at 6 weeks- change at 0 week)/ change at 0 week*100
Time Frame: 0 weeks and 6 weeks
Population: All patients entered into study were analyzed
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Placebo Arm | Vytorin Arm
Number analyzed (Participants) | 10 | 10
percentage of change | 10 (9) | -68 (13)

2. Secondary Outcome: Change in Cream-induced Expression of CD16
Description: Percent change from baseline (0 week) in cream -induced change in CD16 mRNA expression in MNC after 6 weeks of treatment with Vytorin or placebo.
  Outcome calculated as: (change at 6 weeks- change at 0 week)/ change at 0 week*100
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Placebo Arm | Vytorin Arm
Number analyzed (Participants) | 10 | 10
percentage of change | -10 (12) | -57 (13)

3. Secondary Outcome: Change IL-1b mRNA Expression
Description: Percent change from baseline (0 week) in cream -induced change in IL-1b mRNA expression in MNC after 6 weeks of treatment with Vytorin or placebo.
  Outcome calculated as: (change at 6 weeks- change at 0 week)/ change at 0 week*100
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Placebo Arm | Vytorin Arm
Number analyzed (Participants) | 10 | 10
percentage of change | -13 (8) | -74 (15)

4. Secondary Outcome: Change in Plasma Endotoxin (LPS) Concentrations
Description: change from baseline (0 week) in cream -induced change in plasma endotoxin concentration after 6 weeks of treatment with Vytorin or placebo.
  Outcome calculated as: (change at 6 weeks- change at 0 week)
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: EU/ml
Arm/Group | Placebo Arm | Vytorin Arm
Number analyzed (Participants) | 10 | 10
EU/ml | 0.11 (0.09) | -0.23 (0.08)

ADVERSE EVENTS:
Time Frame: 6 WEEKS
Groups:
- Placebo Arm; Vytorin Arm: No Adverse events
Arm/Group | Placebo Arm | Vytorin Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT01420328/Prot_SAP_000.pdf